CLINICAL TRIAL: NCT02977377
Title: Ataksili Hastalarda Tüm Vücut Vibrasyonunun Postüral Kontrol Üzerine Etkileri
Brief Title: The Effects Of Whole Body Vibration On Postural Control In Patients With Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ender AYVAT, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GO 14/397
Record Dates: First submitted 2016-11-18; First posted 2016-11-30 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Ataxia
MeSH Terms: conditions — Ataxia | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole body vibration/ Exercise (Active Comparator): Exercise therapy and whole body vibration will be applied together for 8 weeks. Selected balance, coordination and walking exercises according to the individual needs of patients. Whole body vibration (20-30 Hz, minimum amplitude) will be applied to cases in the form of 4 sets (1 min application and 1min rest) before exercises. After 1 week washout period, exercise program will apply for 8 weeks.
  Interventions: Other: Exercise therapy; Other: Whole body vibration
- Exercise/ Whole body vibration (Active Comparator): Exercise therapy will be applied for 8 weeks. Selected balance, coordination and walking exercises according to the individual needs of patients. After 1 week washout period exercise therapy and whole body vibration will be applied together for 8 weeks.
  Interventions: Other: Exercise therapy; Other: Whole body vibration

INTERVENTIONS:
Other: Exercise therapy — Cases will take the treatment 1-hour, 3 days in a week for 8 weeks.
Other: Whole body vibration — 4 sets, 1 min application and 1min rest whole body vibration and after that exercises. Cases will take the treatment 1-hour, 3 days in a week for 8 weeks.

SUMMARY:
To investigate the effects of whole body vibration on postural control and on the level of satisfaction regarding how to reach the goals of the patients with ataxia

DETAILED DESCRIPTION:
Patients will be randomly assigned to 2 groups, group 1 will take only exercise therapy, group 2 will take exercise therapy and whole body vibration together. After 1 week wash-out period, patients assigned other therapy period. All assessments will be repeated before and after each therapy period. Exercise therapy will consist of selected balance, coordination and walking exercises according to the individual needs of patients. Whole body vibration (20-30 Hz, minimum amplitude) will be applied to cases in the form of 4 sets (1 min application and 1min rest.) Cases will take the treatment 1-hour, 3 days in a week for 8 weeks.

The evaluation parameters consists of demographic information, Computerized Dynamic Posturography, International Cooperative Ataxia Rating Scale, Trunk Impairment Scale, Berg Balance Scale, Barthel Index and Goal Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ataxia
* Ataxic patients who are able to walk 25 m independently

Exclusion Criteria:

* Clinical diagnosis of systemic problems (Diabetes Mellitus, Hypertension)
* Clinical diagnosis of cognitive impairment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Sensory organization test of Computerized Dynamic Posturography (CDP) | change from baseline in sensory component of postural control at 8 weeks
  Computerized Dynamic Posturography (CDP) is a unique assessment technique used to objectively quantify and differentiate among the wide variety of possible sensory, motor, and central adaptive impairments to balance control. CDP has severeal test protocols; a Sensory Organization Test (SOT), Limits of Stability Test (LOS), a Motor Control Test (MCT) and an Adaptation Test (ADT) used in the study. Sensory organization test (SOT) evaluates the relative contributions of vestibular, visual and somatosensory systems to balance maintenance when somatosensory information regarding the orientation of the body's centre of gravity is systematically manipulated.

SECONDARY OUTCOMES:
International Cooperative Ataxia Rating Scale | change from baseline in severity of ataxic symptoms at 8 weeks.
  The ICARS was developed to quantify the level of impairment as a result of ataxia as related to hereditary ataxias. Disorders rated as subscales within the ICARS are: Postural and gait disturbances, Limb Ataxia, Dysarthria and Oculomotor disorders.
Trunk Impairment Scale | change from baseline in impairment of trunk at 8 weeks.
  To measure the motor impairment of the trunk through the evaluation of static and dynamic sitting balance as well as co-ordination of trunk movement. Three subscales: static sitting, balance, dynamic sitting balance and coordination. Each subscale has between three and 10 items.
Berg Balance Scale | change from baseline in balance performance at 8 weeks.
  A 14-item objective measure designed to assess static balance and fall risk. Static and dynamic activities of varying difficulty are performed.Item-level scores range from 0-4, determined by ability to perform the assessed activity. Item scores are summed.Maximum score is 56.
Barthel Index | change from baseline in performance of activitiesof daily living (ADL) at 8 weeks.
  The Barthel includes 10 personal activities. Clinically, the Barthel can be administered via interview, by observation of the patient's performance in a specific setting, or by asking the patient to demonstrate an activity.The response categories of disability in an activity were defined and rated in scale steps (0, 5), (0, 5, 10), (0, 5, 10, 15) dependent on the item. For example, for performance of dressing activity, 0 means dependent, 5 means patient needs help but can do about half unaided, 10 means independent (including buttons, zips, laces, etc.) An overall score is formed by adding scores on each rating. Scores range from 0 (totally dependent) to 100 (fully independent), in steps of 5, with higher scores indicating greater independence.
Goal Assessment Scale | change from baseline in satisfaction regarding how to reach the goals related therapy at 8 weeks.
  The Goal Attainment Scale (GAS) is an individualized outcome measure involving goal selection and goal scaling that is standardized in order to calculated the extent to which a patient's goals are met. Each patient effectively has their own outcome measure, but these measures are scored in a standardized way. "Successful" outcomes are agreed upon prior to intervention. Scoring: Each goal is rated on a 5-point scale. 0 = Patient achieves the expected level; +1 = somewhat more than expected; +2 = much more than expected; -1 = somewhat less than expected; -2 = much less than expected. Overall score is calculated by incorporating the goal outcome scores into a single aggregated T-score. (Optional): Goals may be weighted by the patient for importance or difficulty.
Limits of stability test of Computerized Dynamic Posturography (CDP) | change from baseline in dynamic balance component of postural control at 8 weeks
  Limits of stability test (LOS) assesses dynamic balance during the performance of specific tasks with visual feedback. It quantifies objectively the maximum distance a person can lean in a given direction without losing balance, stepping or reaching for assistance.
Motor Control Test of Computerized Dynamic Posturography (CDP) | change from baseline in automatic motor system component of postural control at 8 weeks
  Motor Control Test (MCT) assesses the ability of the automatic motor system to quickly recover following an unexpected external disturbance. Sequences of platform translations of varied sizes in forward and backward directions elicit automatic postural responses. The size of the translation is scaled to the patient's height to produce sway disturbances of equal size.
Adaptation Test of Computerized Dynamic Posturography (CDP) | change from baseline in postural sway in changes of support surface component of postural control at 8 weeks
  Adaptation Test (ADT) assesses the patient's ability to minimize sway when exposed to irregularities and unexpected changes in support surface properties. Sequences of platform rotations in the toes-up or toes-down direction elicit automatic motor responses.

CONTACTS AND LOCATIONS:
Overall Officials: Ender Ayvat, Msc, Principal Investigator — Hacettepe University; Muhammed Kılınç, Assoc Prof, Principal Investigator — Hacettepe University; Sibel Aksu, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ebersbach G, Edler D, Kaufhold O, Wissel J. Whole body vibration versus conventional physiotherapy to improve balance and gait in Parkinson's disease. Arch Phys Med Rehabil. 2008 Mar;89(3):399-403. doi: 10.1016/j.apmr.2007.09.031. PMID 18295614
- [Result] van Nes IJ, Latour H, Schils F, Meijer R, van Kuijk A, Geurts AC. Long-term effects of 6-week whole-body vibration on balance recovery and activities of daily living in the postacute phase of stroke: a randomized, controlled trial. Stroke. 2006 Sep;37(9):2331-5. doi: 10.1161/01.STR.0000236494.62957.f3. Epub 2006 Aug 10. PMID 16902175
- [Result] Roll JP, Vedel JP, Ribot E. Alteration of proprioceptive messages induced by tendon vibration in man: a microneurographic study. Exp Brain Res. 1989;76(1):213-22. doi: 10.1007/BF00253639. PMID 2753103
- [Result] Torvinen S, Kannus P, Sievanen H, Jarvinen TA, Pasanen M, Kontulainen S, Jarvinen TL, Jarvinen M, Oja P, Vuori I. Effect of four-month vertical whole body vibration on performance and balance. Med Sci Sports Exerc. 2002 Sep;34(9):1523-8. doi: 10.1097/00005768-200209000-00020. PMID 12218749
- [Result] Bruyere O, Wuidart MA, Di Palma E, Gourlay M, Ethgen O, Richy F, Reginster JY. Controlled whole body vibration to decrease fall risk and improve health-related quality of life of nursing home residents. Arch Phys Med Rehabil. 2005 Feb;86(2):303-7. doi: 10.1016/j.apmr.2004.05.019. PMID 15706558
- [Result] Yelnik A, Bonan I. Clinical tools for assessing balance disorders. Neurophysiol Clin. 2008 Dec;38(6):439-45. doi: 10.1016/j.neucli.2008.09.008. Epub 2008 Oct 18. PMID 19026963
- [Result] Trouillas P, Takayanagi T, Hallett M, Currier RD, Subramony SH, Wessel K, Bryer A, Diener HC, Massaquoi S, Gomez CM, Coutinho P, Ben Hamida M, Campanella G, Filla A, Schut L, Timann D, Honnorat J, Nighoghossian N, Manyam B. International Cooperative Ataxia Rating Scale for pharmacological assessment of the cerebellar syndrome. The Ataxia Neuropharmacology Committee of the World Federation of Neurology. J Neurol Sci. 1997 Feb 12;145(2):205-11. doi: 10.1016/s0022-510x(96)00231-6. PMID 9094050
- [Result] Verheyden G, Nieuwboer A, Mertin J, Preger R, Kiekens C, De Weerdt W. The Trunk Impairment Scale: a new tool to measure motor impairment of the trunk after stroke. Clin Rehabil. 2004 May;18(3):326-34. doi: 10.1191/0269215504cr733oa. PMID 15137564
- [Result] Berg KO, Maki BE, Williams JI, Holliday PJ, Wood-Dauphinee SL. Clinical and laboratory measures of postural balance in an elderly population. Arch Phys Med Rehabil. 1992 Nov;73(11):1073-80. PMID 1444775
- [Result] Krasny-Pacini A, Hiebel J, Pauly F, Godon S, Chevignard M. Goal attainment scaling in rehabilitation: a literature-based update. Ann Phys Rehabil Med. 2013 Apr;56(3):212-30. doi: 10.1016/j.rehab.2013.02.002. Epub 2013 Feb 28. PMID 23562111
- [Derived] Ayvat E, Kilinc M, Ayvat F, Onursal Kilinc O, Aksu Yildirim S. The Effect of Whole Body Vibration on Postural Control of Ataxic Patients: a Randomized Controlled Cross-Over Study. Cerebellum. 2021 Aug;20(4):533-541. doi: 10.1007/s12311-021-01233-y. Epub 2021 Jan 21. PMID 33475935